CLINICAL TRIAL: NCT02367027
Title: Single-dose, Open-label, Randomized, 4-way Crossover Study to Compare a Dry Powder Oral Suspension (10 mg and 20 mg Dose of Rivaroxaban) With an Oral Suspension (10 mg of Rivaroxaban) and 10 mg of an Immediate Release Tablet Under Fasting Conditions (10 mg Doses) and Under Fed Conditions (20 mg Dose) in Healthy Male Subjects
Brief Title: Relative Bioavailability Study in Healthy Subjects Comparing 2 Dry Powder Oral Suspensions of Rivaroxaban Under Fasting and 20 mg of an Oral Suspension of Rivaroxaban Under Fed Conditions to 10 mg of an Immediate Release Tablet Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 17769; 2014-004337-69 (EudraCT Number)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Pharmacokinetics
Keywords: Biological Availability; Relative Bioavailability Trial
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 - BAY59-7939 (Experimental): 10 mg oral suspension (dry powder) in fasted conditions
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arn 2 - BAY59-7939 (Experimental): 20 mg oral suspension (dry powder) in fed conditions.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 3 - BAY59-7939 (Experimental): 10 mg oral suspension in fasted conditions
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Arm 4 - BAY59-7939 (Experimental): 10 mg tablet in fasted conditions.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Single dose of 10 mg oral suspension (dry powder) in fasted conditions.
  Arms: Arm 1 - BAY59-7939
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Single dose of 20 mg oral suspension (dry powder) in fed conditions.
  Arms: Arn 2 - BAY59-7939
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Single dose of 10 mg oral suspension in fasted conditions.
  Arms: Arm 3 - BAY59-7939
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Single dose of 10 mg tablet in fasted conditions.
  Arms: Arm 4 - BAY59-7939

SUMMARY:
Rivaroxaban is a substance developed for use in the treatment of blood coagulation disorders.Thrombosis (blood clots) can occur as a result of excessive coagulation activity in the blood vessels. Excessive coagulation activity can occur in children as well, and rivaroxaban is therefore being developed for the treatment of thromboembolic events in children and adolescents. As small children are often unable to swallow tablets, an oral suspension (mixture of a liquid containing finely distributed solids) has been developed which allows dosing according to body weight.The objective of this trial is to compare the bioavailability (proportion of a substance that remains available unchanged in the blood circulation) of a new oral suspension of rivaroxaban with a previously used oral suspension and with a rivaroxaban tablet approved for treatment. In order to evaluate the potential influence of food, the new oral suspension containing 20 mg rivaroxaban will be taken after consuming food. In addition, the pharmacokinetics (concentrations of the drug and breakdown products (metabolites) in blood), safety and tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age: 18 to 55 years (inclusive) at the first screening examination
* White
* Body Mass Index (BMI): ≥18.0 and ≤29.9 kg/m2 at the screening visit.

Exclusion Criteria

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known coagulation disorders (e.g. von Willebrand's disease, hemophilia)
* Known disorders with increased bleeding risk (e.g. periodontosis, hemorrhoids, acute gastritis, peptic ulcer)
* Known sensitivity to common causes of bleeding (e.g. nasal)
* Regular use of medicines and use of medication that may have an impact on the study objectives
* Clinically relevant findings in the ECG such as a second- or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QTc-interval over 450 msec
* Clinically relevant findings in the physical examination
* Clinically relevant deviations of the screened laboratory parameters from reference ranges
* Participation in another clinical study during the preceding 3 months (Last Treatment from previous study to First Treatment of new study)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of rivaroxaban characterized by AUC | Dosing day(15 min, 30 min ,45 min ,1 ,1.5, 2, 2.5 ,3 , 4, 6,8,12,15 hours), at 48 hr after administration), at 72 hr after administration)
  AUC:area under the concentration vs. time curve from zero to infinity after single (first) dose
Plasma concentration of rivaroxaban characterized by AUC/D | Dosing day(15 min, 30 min ,45 min ,1 ,1.5, 2, 2.5 ,3 , 4, 6,8,12,15 hours),at 48 hr after administration),at 72 hr after administration)
  AUC/D: AUC divided by dose
Plasma concentration of rivaroxaban characterized by Cmax | Dosing day(15 min, 30 min ,45 min ,1 ,1.5, 2, 2.5 ,3 , 4, 6,8,12,15 hours),at 48 hr after administration),at 72 hr after administration)
  Cmax: maximum drug concentration in plasma after single dose administration
Plasma concentration of rivaroxaban characterized by Cmax/D | Dosing day(15 min, 30 min ,45 min ,1 ,1.5, 2, 2.5 ,3 , 4, 6,8,12,15 hours),at 48 hr after administration),at 72 hr after administration)
  Cmax/D: Cmax divided by dose

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mannheim, Baden-Wurttemberg, Germany